CLINICAL TRIAL: NCT00255827
Title: A Phase I/II Study of Algenpantucel-L (HyperAcute Pancreas) an Antitumor Vaccination Using Alpha(1,3)Galactosyltransferase Expressing Allogeneic Tumor Cells in Patients With Pancreatic Cancer
Brief Title: Vaccine Treatment for Surgically Resected Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Nicholas N. Vahanian, M.D., Chief Medical and Operations Officer, NewLink Genetics Corporation
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG0105
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Algenpantucel-L

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: HyperAcute-Pancreatic Cancer Vaccine

SUMMARY:
This 2-phase study will determine the safety of treating patients with pancreatic cancer with the genetically engineered HyperAcute-Pancreatic cancer vaccine. It will establish the proper vaccine dose and will examine side effects and potential benefits of the treatment. The vaccine contains killed pancreatic cancer cells containing a mouse gene that causes the production of a foreign pattern of protein-sugars on the cell surface. It is hoped that the immune response to the foreign substance will stimulate the immune system to attack the patient's own cancer cells that have similar proteins without this sugar pattern, causing the tumor to remain stable or shrink.

Patients 18 years of age or older with pancreatic cancer that has been surgically resected may be eligible for this study. Candidates will be screened with medical history and physical examination, blood tests, urinalysis, chest x-rays and CT scans. MRI, PET, and ultrasound scans may be obtained if needed.

Participants will receive twelve vaccinations two weeks apart from each other. The vaccines will be injected under the skin, similar to the way a tuberculosis skin test is given. Phase I of the study will treat successive groups of patients with increasing numbers of the vaccine cells to evaluate side effects of the treatment and determine the optimum dose. Phase II will look for any beneficial effects of the vaccine given at the highest dose found to be safe in Phase I. Monthly blood samples will be drawn during the 6 months of vaccine treatment. In addition, patient follow-up visits will be scheduled every 2 months for the remaining first year (6 months) after vaccination and then every 3 months for the next 2 years for the following tests and procedures to evaluate treatment response and side effects:

Medical history and physical examination Blood tests X-rays and various scans (nuclear medicine/CT/MRI) FACT-Hep Assessment questionnaire to measure the impact of treatment on the patient's general well-being. The questionnaire is administered before beginning treatment, monthly during treatment, and during follow-up visits after completing the treatment. It includes questions on the severity of pancreatic cancer symptoms and the ability to perform normal activities of daily life.

DETAILED DESCRIPTION:
According to statistics of the American Cancer Society, an estimated 31,000 individuals will be diagnosed with pancreatic cancer and 25,000 will die of the disease, making it the fifth leading cause of U.S. cancer deaths this year despite all current therapy. This protocol attempts to exploit an approach to pancreatic cancer immunotherapy using a naturally occurring barrier to xenotransplantation in humans in an attempt to vaccinate patients against their pancreatic cancer. The expression of the murine alpha (1,3) galactosyltransferase [alpha (1,3) GT] gene results in the cell surface expression of alpha (1,3) galactosyl-epitopes (alpha-gal) on membrane glycoproteins and glycolipids. These epitopes are the major target of the hyperacute rejection response that occurs when organs are transplanted from non-primate donor species into man. Human hosts often have pre-existing anti-alpha-gal antibodies that bind alpha-gal epitopes and lead to rapid activation of complement and cell lysis. The pre-existing anti-alpha-gal antibodies found in most individuals are thought to be due to exposure to alpha-gal epitopes that are naturally expressed on normal gut flora leading to chronic immunological stimulation. These antibodies may comprise up to 1% of serum IgG. In this Phase I/II trial, patients with surgically resected pancreatic cancer will undergo a series of twelve intradermal injections with a vaccine composed of irradiated allogeneic pancreatic cancer cell lines (HAPa-1 and HAPa-2) that have been transduced with a recombinant Moloney murine leukemia virus (MoMLV)-based retroviral vector expressing the murine alpha (1,3) GT gene. Endpoints of the study include determination of dose-limiting toxicity (DLT), maximum tolerated dose (MTD), tumor and immunological responses.

ELIGIBILITY:
Inclusion Criteria:

* A histological diagnosis of adenocarcinoma or other exocrine carcinoma of the pancreas. The patient's pathology must be reviewed and confirmed by Northwestern University's Pathology Department.
* AJCC Stage I or II Pancreatic carcinoma. Patients must have undergone surgical resection for the tumor.
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 2.
* Serum albumin greater than or equal to 2.5 gm/dL.
* Expected survival greater than or equal to 6 months.
* Subjects must have a negative serology for Hep B, C and HIV prior to entering study.
* All On-Study Tests must be less than or equal to Grade I toxicity for patient to be eligible for study, excluding serum LDH levels. PT, PTT must be less than or equal to 1.5 x ULN except for patients who are on therapeutic anticoagulant therapy.
* Adequate organ function including:

Marrow: hemoglobin greater than or equal to 10.0 gm/dL, absolute granulocyte count (AGC) greater than or equal to 1500/mm3, platelets greater than or equal to 100,000/mm3, absolute lymphocyte count greater than or equal to 475/mm3.

Hepatic: serum total bilirubin less than or equal to 1.5 x ULN mg/dL, ALT (SGPT) and AST (SGOT) less than or equal to 2.5 x upper limit of normal (ULN).

Renal: serum creatinine (sCr) less than or equal to 2.0 x ULN, or creatinine clearance (Ccr) greater than or equal to 30 mL/min.

* Prior therapy for pancreatic cancer that may include surgery and/or different neoadjuvant chemotherapy or adjuvant chemo-radiation regimens, or radiation therapy. Patients who undergo surgical resection and refuse chemotherapy or radiation therapy will be eligible.
* Patients must be greater than or equal to 4 weeks since surgery if treated with neoadjuvant therapy or greater than or equal to 4 weeks since conclusion of chemo-radiation if treated with post-operative adjuvant therapy and recovered from the toxicity of prior treatment to less than or equal to Grade I, exclusive of alopecia or fatigue.
* Patients must have the ability to understand the study, its inherent risks, side effects and potential benefits and be able give written informed consent to participate. Patients may not be consented by a durable power of attorney (DPA).
* All subjects of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental product, and for one month after the last immunization.

Exclusion Criteria:

* Age <18-years-old.
* Active metastases.
* Hypercalcemia > 2.9 mmol/L, unresponsive to standard therapy (e.g., I.V. hydration, diuretics, calcitonin or bisphosphonate therapy).
* Other malignancy within five years, unless the probability of recurrence of the prior malignancy is <5%. Patient's curatively treated for squamous and basal cell carcinoma of the skin or patients with a history of malignant tumor in the past that have been disease free for at least five years are also eligible for this study.
* History of organ transplant or current active immunosuppressive therapy (such as cyclosporine, tacrolimus, etc.).
* Subjects taking systemic corticosteroid therapy for any reason are not eligible. Subjects receiving inhaled or topical corticosteroids are eligible. Subjects who require systemic corticosteroids after beginning vaccination, will be removed from study.
* Significant or uncontrolled congestive heart failure (CHF), myocardial infarction or significant ventricular arrhythmias within the last six months.
* Active infection or antibiotics within 1-week prior to study, including unexplained fever (temp > 38.1C).
* Autoimmune disease (e.g., systemic lupus erythematosis (SLE), rheumatoid arthritis (RA), etc.). Patients with a remote history of asthma or mild active asthma are eligible.
* Other serious medical conditions that may be expected to limit life expectancy to less than 2 years (e.g., liver cirrhosis) or a serious illness in medical opinion of the clinical investigator.
* Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc.).
* A known allergy to any component of the alpha(1,3)galactosyltransferase tumor vaccine or cell lines.
* Prior splenectomy.
* Pregnant or nursing women due to the unknown effects of vaccination on the developing fetus or newborn infant. (For patients with child bearing potential, a βHCG must be completed within 7 days of first vaccination).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To assess the side effects, dose-limiting toxicity and maximum tolerated dose. | 6 months

SECONDARY OUTCOMES:
To assess the rate of recurrence after treatment. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mulcahy, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States